CLINICAL TRIAL: NCT00847821
Title: RNA Expression Analysis Of Endometrial Biopsies Comparing Placebo, Bazedoxifene/ Conjugated Estrogens And Raloxifene
Brief Title: Observational Study Analyzing RNA Expression Of Endometrial Biopsy Samples From Placebo, Bazedoxifene/Conjugated Estrogens And Raloxifene
Status: Terminated | Type: Observational
Why Stopped: See termination reason in detailed description.
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc
Other Study IDs: 3115A1-1125; B2311003
Record Dates: First submitted 2009-02-18; First posted 2009-02-19 (Estimated); Last update posted 2010-09-06 (Estimated); Status verified 2010-09

CONDITIONS: Postmenopause
MeSH Terms: interventions — bazedoxifene; Raloxifene Hydrochloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Endometrial biopsy blocks
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (8):
- Bazedoxifene 10 mg/CE 0.625 mg
  Interventions: Drug: Bazedoxifene 10 mg/CE 0.625 mg
- Bazedoxifene 20 mg/CE 0.625 mg
  Interventions: Drug: Bazedoxifene 20 mg/CE 0.625 mg
- Bazedoxifene 40 mg/CE 0.625 mg
  Interventions: Drug: Bazedoxifene 40 mg/CE 0.625 mg
- Bazedoxifene 10 mg/CE 0.45 mg
  Interventions: Drug: Bazedoxifene 10 mg/CE 0.45 mg
- Bazedoxifene 20 mg/CE 0.45 mg
  Interventions: Drug: Bazedoxifene 20 mg/CE 0.45 mg
- Bazedoxifene 40 mg/CE 0.45 mg
  Interventions: Drug: Bazedoxifene 40 mg/CE 0.45 mg
- Raloxifene 60 mg
  Interventions: Drug: Raloxifene 60 mg
- Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bazedoxifene 10 mg/CE 0.625 mg — No dose taken during this study; however, this intervention was taken while study 3115A1-303 was ongoing. In the 3115A1-303 study, test article was supplied as bazedoxifene/CE tablets in capsules. The dosage was one capsule orally, once daily, at approximately the same time each day on a continuous regiment for 2 years, or until early discontinuation from the study.
  Groups: Bazedoxifene 10 mg/CE 0.625 mg
Drug: Bazedoxifene 20 mg/CE 0.625 mg — No dose taken during this study; however, this intervention was taken while study 3115A1-303 was ongoing. In the 3115A1-303 study, test article was supplied as bazedoxifene/CE tablets in capsules. The dosage was one capsule orally, once daily, at approximately the same time each day on a continuous regiment for 2 years, or until early discontinuation from the study.
  Groups: Bazedoxifene 20 mg/CE 0.625 mg
Drug: Bazedoxifene 40 mg/CE 0.625 mg — No dose taken during this study; however, this intervention was taken while study 3115A1-303 was ongoing. In the 3115A1-303 study, test article was supplied as bazedoxifene/CE tablets in capsules. The dosage was one capsule orally, once daily, at approximately the same time each day on a continuous regiment for 2 years, or until early discontinuation from the study.
  Groups: Bazedoxifene 40 mg/CE 0.625 mg
Drug: Bazedoxifene 10 mg/CE 0.45 mg — No dose taken during this study; however, this intervention was taken while study 3115A1-303 was ongoing. In the 3115A1-303 study, test article was supplied as bazedoxifene/CE tablets in capsules. The dosage was one capsule orally, once daily, at approximately the same time each day on a continuous regiment for 2 years, or until early discontinuation from the study.
  Groups: Bazedoxifene 10 mg/CE 0.45 mg
Drug: Bazedoxifene 20 mg/CE 0.45 mg — No dose taken during this study; however, this intervention was taken while study 3115A1-303 was ongoing. In the 3115A1-303 study, test article was supplied as bazedoxifene/CE tablets in capsules. The dosage was one capsule orally, once daily, at approximately the same time each day on a continuous regiment for 2 years, or until early discontinuation from the study.
  Groups: Bazedoxifene 20 mg/CE 0.45 mg
Drug: Bazedoxifene 40 mg/CE 0.45 mg — No dose taken during this study; however, this intervention was taken while study 3115A1-303 was ongoing. In the 3115A1-303 study, test article was supplied as bazedoxifene/CE tablets in capsules. The dosage was one capsule orally, once daily, at approximately the same time each day on a continuous regiment for 2 years, or until early discontinuation from the study.
  Groups: Bazedoxifene 40 mg/CE 0.45 mg
Drug: Raloxifene 60 mg — No dose taken during this study; however, this intervention was taken while study 3115A1-303 was ongoing. In the 3115A1-303 study, test article was supplied as raloxifene tablets in capsules. The dosage was one capsule orally, once daily, at approximately the same time each day on a continuous regiment for 2 years, or until early discontinuation from the study.
  Groups: Raloxifene 60 mg
Drug: Placebo — No dose taken during this study; however, this intervention was taken while study 3115A1-303 was ongoing. In the 3115A1-303 study, test article was supplied as placebo capsules. The dosage was one capsule orally, once daily, at approximately the same time each day on a continuous regiment for 2 years, or until early discontinuation from the study.
  Groups: Placebo

SUMMARY:
This study is an observational study analyzing the biopsy samples collected from subjects that participated in Study 3115A1-303 (NCT00675688). These endometrial biopsy samples will be de-identified at an anatomical laboratory and then sent to a molecular biology lab where an RNA extraction and analysis will be performed. The purpose of this study is to compare specific endometrial gene regulation at the level of mRNA expression in samples from placebo, bazedoxifene/conjugated estrogens, and raloxifene treated groups with a known set of genes that have been previously identified to be associated with estrogenization, endometrial hyperplasia, and endometrial cancer.

DETAILED DESCRIPTION:
The termination date was June 23, 2010. The study was terminated because the endometrial biopsy blocks from the 3115A1-303 study that were to be used for this study need to be retained and accessible in case of a regulatory inspection of the 303 protocol. Additionally, the Brazilian sites were not likely not to receive national IRB (CONEP) approval, and enrollment could not be met without the inclusion of these subjects. The study was not terminated due to safety concerns.

ELIGIBILITY:
Inclusion Criteria:

* Each subject must have participated in study 3115A1-303 and must have satisfied all of the following criteria:
* Has completed 24 months of treatment.
* Was at least 80% compliant with study drug administration.

Exclusion Criteria:

* Endometrial biopsy at baseline, month 6 or month 24 that were technically unacceptable
* Did not have an endometrial biopsy at all of the required timepoints (baseline, month 6, month 24)

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postmenopausal women who participated in and completed the 3115A1-303 study, were at least 80% compliant with test article administration during the study, and have provided a new signed and written informed consent for study 3115A1-1125.
Sampling Method: Non-Probability Sample
Enrollment: 185 (Actual)
Dates: Start 2009-05; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Endometrial gene regulation at the level of mRNA expression in placebo, Bazedoxifene/CE, and raloxifene treated groups | Baseline, 6 months and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (22):
- United States (22):
  - Pfizer Investigational Site, Fort Myers, Florida
  - Pfizer Investigational Site, Gainesville, Florida
  - Pfizer Investigational Site, New Port Richey, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Decatur, Georgia
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Southfield, Michigan
  - Pfizer Investigational Site, Chaska, Minnesota
  - Pfizer Investigational Site, Billings, Montana
  - Pfizer Investigational Site, New Brunswick, New Jersey
  - Pfizer Investigational Site, Las Vegas, New Mexico
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Wexford, Pennsylvania
  - Pfizer Investigational Site, Greenville, South Carolina
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Charlottesville, Virginia
  - Pfizer Investigational Site, Norfolk, Virginia

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3115A1-1125&StudyName=Observational%20Study%20Analyzing%20RNA%20Expression%20Of%20Endometrial%20Biopsy%20Samples%20From%20Placebo%2C%20Bazedoxifene/Conjugated%20Estrogens%20And%20Raloxifene